CLINICAL TRIAL: NCT03129529
Title: Comparing the Effect of Focused and Radial Extracorporeal Shock Waves on Post-stroke Hypertonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Gwo-Chi Hu,PHD, PHD, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15MMHIS194e
Record Dates: First submitted 2017-04-20; First posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No

ARMS (2):
- focused shock wave (Experimental): Treatment was administered directly to the middle of muscle bellies of the spastic triceps surae muscle in three sessions, with one week interval. During each session, 3000 pulses (1500 shots in the gastrocnemius and 1500 shots in the soleus muscle) were delivered at 5 Hz. The intensities of FSWT were 0.10 mJ/mm2.
  Interventions: Device: Focused shock wave
- radial shock wave (Experimental): Treatment was administered directly to the middle of muscle bellies of the spastic triceps surae muscle in three sessions, with one week interval. During each session, 3000 pulses (1500 shots in the gastrocnemius and 1500 shots in the soleus muscle) were delivered at 5 Hz.The intensities of RSWT were 2.0 bar.
  Interventions: Device: Radial shock wave

INTERVENTIONS:
Device: Focused shock wave — The outcome evaluation include ankle range of motion (ROM), modified Ashworth scale (MAS),modified Tardieu scale (MTS), baropodometric measurement, and gait speed.
  Arms: focused shock wave
Device: Radial shock wave — The outcome evaluation include ankle range of motion (ROM), modified Ashworth scale (MAS),modified Tardieu scale (MTS), baropodometric measurement, and gait speed.
  Arms: radial shock wave

SUMMARY:
The main purpose of this study is to compare treatment efficacy of focused and radial extracorporeal shock waves on spasticity in chronic stroke patient

DETAILED DESCRIPTION:
This study is a prospective and double-blinded randomized control trial. Thirty-two stroke patients with spastic equinus were randomly assigned to receive three sessions of either focused shockwave therapy or radial shockwave therapy at 1-week intervals. The intensities that were used during FSWT (0.1 mJ/mm2) and RSWT (2 bar) were comparable. Patients were evaluated at baseline and at 1, 4, 8 weeks after the final shockwave treatment. The primary outcome measure was modified Ashworth scale (MAS) score. Secondary outcome measures were Tardieu scale, ankle passive range of motion, plantar contact area during gait, and gait speed. A linear mixed model with repeated measures was used to compare each outcome measure between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* aged greater than 18 years old;
* at least 6 months since onset of last stroke;
* triceps surae muscle tone graded at least 1+ on the Modified Ashworth Scale (MAS) score;
* ability to walk alone with/without orthosis.

Exclusion Criteria:

* Exclusion criteria included fixed ankle joint contracture, previous treatment of the affected leg with neurolytic or surgical procedures, concomitant progressive central nervous system diseases, and skin breakdown, vascular disease in the affected leg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline of spasticity on 1st, 4th, 8th weeks after treatment. | 1, 4, 8 week
  Using the modyfied Ashworth Scale to measure the spasticity before treatment and multiple time frame after treatment.

SECONDARY OUTCOMES:
Change from baseline of range of motion on 1st, 4th, 8th weeks after treatment. | 1, 4, 8 week
  Using the digital goniometer to measure the passive range of motion before treatment and multiple time frame after treatment.
Change from baseline of modified Tardieu scale on 1st, 4th, 8th weeks after treatment. | 1, 4, 8 week
  Using the modified Tardieu scale (MTS) to measure the spasticity before treatment and multiple time frame after treatment.
Change from baseline of foot contact area on 1st, 4th, 8th weeks after treatment. | 1, 4, 8 week
  Using the baropodometric measurement to measure the foot contact area before treatment and multiple time frame after treatment.
Change from baseline of gait speed on 8th weeks after treatment. | 8 week
  Using the 10 meters walking test to measure the gait speed before treatment and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan